CLINICAL TRIAL: NCT06599450
Title: Clinical and Radiographic Comparison of Symphyseal and Parasymphyseal Single Implant Versus Two Implants in Complete Mandibular Overdentures
Brief Title: Single vs. Two Implants for Mandibular Overdentures
Acronym: SIMO/TIMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Ezzat Ahmed Al-Gazzar, Principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUAREC20210006-5
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bleeding on Probing; Alveolar Bone Loss; Mastication; Dental Plaque; Periodontal Index
MeSH Terms: conditions — Alveolar Bone Loss; Dental Plaque

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One median implant (Active Comparator): One median implant to retain mandibular complete overdenture
  Interventions: Device: Root form dental implant
- One parasymphyseal implant (Active Comparator): One parasymphyseal implant to retain mandibular complete overdenture
  Interventions: Device: Root form dental implant
- Two implants (Active Comparator): Two implants in the intraforaminal distance to retain mandibular complete overdenture
  Interventions: Device: Root form dental implant

INTERVENTIONS:
Device: Root form dental implant — Placement of titanium endosteal root form threaded tapered two-piece dental implant to assist mandibular complete overdenture

SUMMARY:
This study aimed to compare the use of single implants in the symphyseal and parasymphyseal, and two implants were inserted in the canine area bilaterally to assist mandibular complete overdentures regarding clinical evaluation, marginal bone loss, and masticatory efficiency. The null hypothesis was that there was no statistically significant difference in clinical evaluation, marginal bone loss, and masticatory efficiency among single symphyseal implants, single parasymphyseal implants, and two-implant-assisted complete mandibular overdentures.

DETAILED DESCRIPTION:
This randomized, controlled clinical trial compared the symphyseal and parasymphyseal single implants versus two implants in complete mandibular overdentures. Fifteen completely edentulous male patients (50-65 years) were chosen and randomly grouped into three equal groups (five patients in each) according to the position and number of the received implants to assist mandibular complete overdentures. Group I: single median implant. Group II: single parasymphyseal implant. Group III: two implants were inserted in the canine area bilaterally. After three months of osseointegration, the lower denture was transformed into an implant-assisted complete mandibular overdenture. Clinical observations were documented on the day of loading, three, six, and nine months later for each implant. Follow-up CBCT scans were performed to assess marginal bone loss on the day of loading, six and twelve months later. The masticatory efficiency evaluation was conducted one month and three months after loading.

ELIGIBILITY:
Inclusion Criteria:

* patients with a class I Maxillo-mandibular jaw relationship
* patients with residual ridges had normal morphology, were free from severe bony undercuts or flabby tissue, and were covered by firm mucoperiosteum.
* A cone beam CT of the lower arch was made to detect the presence of pathological lesions, remaining roots, or impacted teeth in the arch and evaluate both bone quality and quantity, especially in the area of interest

Exclusion Criteria:

* patients with current chemotherapy or radiotherapy, bleeding disorders, uncontrolled diabetes
* patients with a history of drug therapy that interferes with bone resorption or deposition (e.g., the prolonged use of glucocorticoids, antiresorptive medications, selective serotonin reuptake inhibitors, and proton-pump inhibitors),
* Those with any physical reasons that could affect follow-up, psychiatric problems, heavy smokers, drug or alcohol addicts, immunocompromised patients, abnormal jaw relationship, inadequate inter arch space.
* patients with temporomandibular disorders and para-functional habits (e.g., bruxing and clenching).

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Change in the plaque index | The plaque index was documented at follow-up visits on the day of loading, three, six, and nine months later for each implant.
  The presence and amount of plaque were determined at the four sites around the implant (mesial, distal, buccal, and lingual) and scored from zero to three. Grade 0: No plaque by probing. Grade 1: film of plaque detected by probing. Grade 2: Visible plaque with the naked eye. Grade 3: abundant soft material in the sulcus, mucosal margin, and adjacent implant surface.
Change in the pocket depth | The pocket depth was documented at follow-up visits on the day of loading, three, six, and nine months later for each implant.
  The pocket depth was measured by inserting a graduated plastic periodontal probe between the oral sulcular epithelium and the implant with minimal pressure at the midpoint of the four surfaces. The distance from the bottom of the sulcus to the mucosal margin was measured and recorded to the nearest millimeter; the mean of four readings was considered the pocket depth for this group at the chosen time
Change in the bleeding index | The bleeding index was documented at follow-up visits on the day of loading, three, six, and nine months later for each implant.
  The bleeding index was assessed for the four surfaces while measuring the pocket depth if the bleeding was visible after probing within 20 seconds. It is typically scored as 0 (no bleeding), 1 (bleeding point), 2 (single line of blood), or 3 (heavy or profuse bleeding). The mean of four readings was considered the bleeding index for this group at the chosen time
Change in bone level around implant | Immediately after loading, six months, and twelve months later
  Calculating average bone height involves dividing the sum of buccal, lingual, mesial, and distal bone height by 4. The real bone loss can be calculated by subtraction from the implant length
Change in the masticatory efficiency | The masticatory efficiency was documented at follow-up visits one month and three months after the overdenture insertion
  The masticatory efficiency was assessed when the patient ate three different types of food (carrot, apple, and banana) with varying degrees of hardness, cut into standardized pieces (1 cm cube each). The collected data included the following measurements: the chewing stroke count before the first swallow, the chewing stroke count until the oral cavity is empty of food, the count of swallows until the oral cavity is empty of food, the time estimated in seconds until the first swallow, and the time estimated in seconds until the oral cavity is empty of food.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed B El-okl, Professor, Study Chair — Removable Prosthodontics, Al-Azhar University, Asuit, EGY
Locations (1):
- Faculty of Dental Medicine, Al-Azhar University, Assuit, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No